CLINICAL TRIAL: NCT02653547
Title: Influence of Treatment Duration and Stimulation Frequency on Repetitive Transcranial Magnetic Stimulation in Chronic Tinnitus
Brief Title: Influence of Treatment Duration and Stimulation Frequency on rTMS in Chronic Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., M.D., Ph.D., University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: dur-freq-rTMS-tin
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Chronic Tinnitus
Keywords: tinnitus; transcranial random noise stimulation; rTMS; multisite stimulation; non-invasive brain stimulation
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- standard multisite four weeks (Experimental): Combined high-frequency dorsolateral prefrontal (unilateral) and low frequency temporoparietal (bilateral) stimulation; complete treatment of four weeks
  Interventions: Other: standard multisite four weeks
- high-frequency multisite four weeks (Experimental): Combined high-frequency dorsolateral prefrontal (unilateral) and high-frequency temporoparietal (bilateral) stimulation; complete treatment of four weeks
  Interventions: Other: high-frequency multisite four weeks
- standard multisite two weeks (Experimental): Combined high-frequency dorsolateral prefrontal (unilateral) and low frequency temporoparietal (bilateral) stimulation; discontinuation after two weeks
  Interventions: Other: standard multisite two weeks
- high-frequency multisite two weeks (Experimental): Combined high-frequency dorsolateral prefrontal (unilateral) and high-frequency temporoparietal (bilateral) stimulation; discontinuation after two weeks
  Interventions: Other: high-frequency multisite two weeks

INTERVENTIONS:
Other: standard multisite four weeks — Repetitive transcranial magnetic stimulation (Magventure): 1000 stimuli of 20 Hz rTMS over the left DLPFC (110% motor threshold) followed by 1000 stimuli of 1 Hz rTMS over the left temporoparietal cortex (110% motor threshold) followed by 1000 stimuli of 1 Hz rTMS over right temporoparietal cortex (110% motor threshold). Patients continue treatment after two weeks for further two weeks of treatment (20 treatment days).
  Arms: standard multisite four weeks
Other: high-frequency multisite four weeks — Repetitive transcranial magnetic stimulation (Magventure): 1000 stimuli of 20 Hz rTMS over the left DLPFC (110% motor threshold) followed by 1000 stimuli of 20 Hz rTMS over the left temporoparietal cortex (110% motor threshold) followed by 1000 stimuli of 20 Hz rTMS over right temporoparietal cortex (110% motor threshold). Patients continue treatment after two weeks for further two weeks of treatment (20 treatment days).
  Arms: high-frequency multisite four weeks
Other: standard multisite two weeks — Repetitive transcranial magnetic stimulation (Magventure): 1000 stimuli of 20 Hz rTMS over the left DLPFC (110% motor threshold) followed by 1000 stimuli of 1 Hz rTMS over the left temporoparietal cortex (110% motor threshold) followed by 1000 stimuli of 1 Hz rTMS over right temporoparietal cortex (110% motor threshold). Patients discontinue treatment after two weeks (10 treatment days).
  Arms: standard multisite two weeks
Other: high-frequency multisite two weeks — Repetitive transcranial magnetic stimulation (Magventure): 1000 stimuli of 20 Hz rTMS over the left DLPFC (110% motor threshold) followed by 1000 stimuli of 20 Hz rTMS over the left temporoparietal cortex (110% motor threshold) followed by 1000 stimuli of 20 Hz rTMS over right temporoparietal cortex (110% motor threshold). Patients discontinue treatment after two weeks (10 treatment days).
  Arms: high-frequency multisite two weeks

SUMMARY:
Patients receive two weeks of treatment (prefrontal high-frequency and bilateral low-frequency rTMS vs. prefrontal high-frequency and bilateral high-frequency rTMS). After two weeks of treatment they can decide if they want to quit the treatment or if they want to proceed with the treatment for another two weeks.

DETAILED DESCRIPTION:
Tinnitus is the phantom auditory perception of sound in the absence of an external or internal acoustic stimulus. It is a frequent problem which can interfere significantly with the ability to lead a normal life. Tinnitus has been shown to be generated in the brain, as a result of functional reorganization of auditory and non-auditory neural pathways. Low-frequency repetitive transcranial magnetic stimulation (rTMS) applied to the temporoparietal areas has been investigated for the treatment of tinnitus based on the rationale to reduce increased activity of the auditory system. Furthermore, high-frequency stimulation of the left frontal cortex was added to this standard treatment based on rTMS studies in affective disorders and the association of tinnitus distress with depressivity. Thus, high-frequency stimulation of the left prefrontal cortex and low-frequency stimulation of bilateral temporoparietal cortex was introduced as new treatment scheme in chronic tinnitus (multisite standard).

Additionally, there is also evidence that high-frequency stimulation of the temporoparietal cortex is effective in chronic tinnitus. Furthermore, standard treatment in chronic tinnitus is two weeks (ten treatment days) which is shorter than the standard in rTMS in affective disorders. Thus, the aim of the present trial is to investigate the influence of high-frequency stimulation of the temporoparietal cortex and of increasing the number of treatment days.

Patients receive two weeks of treatment (prefrontal high-frequency and bilateral low-frequency rTMS vs. prefrontal high-frequency and bilateral high-frequency rTMS). After two weeks of treatment they can decide if they want to quit the treatment or if they want to proceed with the treatment for another two weeks.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* duration of tinnitus more than 6 months
* bothersome chronic tinnitus

Exclusion Criteria:

* not stable internal, mental, and neurological diseases
* contraindication for rTMS (pacemaker, metal implants, pregnancy, epilepsy, status post severe craniocerebral injury )
* uninvolvement in other treatment studies for tinnitus at the same time

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-01; Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
change in tinnitus questionnaire | week12
  change in tinnitus questionnaire

SECONDARY OUTCOMES:
change in tinnitus questionnaire | week2, week3, week4, week12
  change in tinnitus questionnaire
change in tinnitus handicap inventory | week2, week3, week4, week12
  change in tinnitus handicap inventory
change in tinnitus numeric rating scales | week2, week3, week4, week12
  change in tinnitus numeric rating scales
change in major depression inventory | week2, week3, week4, week12
  change in major depression inventory
change in clinical global impression | week2, week3, week4, week12
  change in clinical global impression
change in quality of life | week2, week3, week4, week12
  change in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, Principal Investigator — University of Regensburg, Department of Psychiatry
Locations (1):
- University of Regensburg- Dept of Psychiatry, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided